CLINICAL TRIAL: NCT04982510
Title: Retention of 3D Printed Bases Using Prefabricated Thermoplastic Trays and Conventional Custom Impression Trays: Randomized Controlled Trial
Brief Title: Accuracy of 3D Printed Complete Dentures Using Two Impression Techniques: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sonal Abdelbaseer, Principal investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4421
Record Dates: First submitted 2021-07-15; First posted 2021-07-29 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Edentulism Nos
Keywords: digital dentures, definitive impression, thermoplastic trays, printed denture, 3D, rapid prototyping
MeSH Terms: interventions — Denture, Complete

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermoplastic tray definitive impression (Experimental)
  Interventions: Device: complete denture
- Conventional tray definitive impression (Active Comparator)
  Interventions: Device: complete denture

INTERVENTIONS:
Device: complete denture — 3D printed complete denture

SUMMARY:
the aim of this crossover randomized controlled clinical trial is comparing retention of 3D printed maxillary complete dentures produced from thermoplastic impression trays and conventional acrylic impression trays.

The research hypothesis is that there is no difference in patient satisfaction and retention of dentures constructed from definitive impression using the conventional tray and the prefabricated thermoplastic tray

ELIGIBILITY:
Inclusion Criteria:

* Male edentulous patients.
* Cooperative and highly motivated patients.
* Patients with well or moderately developed ridges and healthy attached mucosa of appropriate thickness free from inflammation

Exclusion Criteria:

* Patients with recent extraction less than 3 months ago
* Patients with Parkinson's disease
* Patients with xerostomia.
* Patients with allergy to resins.
* Pathological changes of residual ridges.
* Patient with sever undercuts, or irregular bony exostosis.
* Patients with flabby and flat ridges.
* Patients with medical or psychological conditions that hinder co-operation.
* Patients with class II or III jaw relation.

Max Age: 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Maxillary complete denture base retention | 2 weeks after denture insertion
  A loop will be attached to each denture base at the position of geographic center using self cure acrylic resin and the retention will be measured by applying the forces perpendicular to the denture using Digital Force Meter Each base will be tested 3 times and the average will be calculated.

SECONDARY OUTCOMES:
Patient satisfaction | 2 weeks
  patient satisfaction data will be collected through questionnaire and graded by Visual analogue scale for both study arms

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided